CLINICAL TRIAL: NCT02210819
Title: XALIA LEA- Xarelto for Long-term and Initial Anticoagulation in Venous Thromboembolism (VTE) in Latin America, EMEA and Asia
Brief Title: Treatment of Venous Thromboembolism (VTE) With Either Rivaroxaban or Current Standard of Care Therapy
Acronym: XALIA LEA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17237; XA1402 (Other: Company internal)
Record Dates: First submitted 2014-05-20; First posted 2014-08-07 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE)
Keywords: Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban: Patients who will be treated for an acute venous thromboembolism (VTE) with rivaroxaban.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Standard of care: Patients who will be treated for an acute venous thromboembolism (VTE) with current standard of care.
  Interventions: Drug: Recommended VTE pharmacological treatments according to international guidelines

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Cohort participants are classified as "rivaroxaban" patient, if the patient receives initial rivaroxaban VTE treatment. Dosing according to daily clinical routine
  Groups: Rivaroxaban
Drug: Recommended VTE pharmacological treatments according to international guidelines — Cohort participants are classified as "Standard of care" patients, if the patient receives recommended VTE pharmacological treatments according to international guidelines, e.g. unfractionated heparin, LMWH, fondaparinux, VKA, if these are also approved pharmacological treatments for VTE in the respective country. Dosing according to daily clinical routine.
  Groups: Standard of care

SUMMARY:
Following the findings of the clinical trials in drug development, this global non-interventional cohort field study will investigate rivaroxaban under clinical practice conditions in comparison with current standard of care for patients with acute venous thoromboembolism (VTE).

The main goal is to analyze long-term safety in the use of rivaroxaban in the treatment of acute VTE in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, who are at >=18 years
* Diagnosis of acute DVT and/or PE, objectively confirmed
* Indication for anticoagulation therapy for at least 12 weeks
* Willing to participate in this study and available for follow-up

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- and outpatients in sites participating in the study.
Sampling Method: Probability Sample
Enrollment: 1987 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Number of major bleedings defined as overt bleeding | Up to 2 years
  Major bleedings defined as overt bleeding are associated with: A fall in hemoglobin of ≥2 g/dL; or a transfusion of ≥2 units of packed red blood cells or whole blood; or occurrence at a critical site
Number of patients with symptomatic recurrent venous thromboembolic events | Up to 2 years
All cause mortality | Up to 2 years

SECONDARY OUTCOMES:
Number of adverse cardiovascular events | Up to 2 years
  Number of cardiovascular events will be used for descriptive statistics to summarize safety variables.
Number of patients with other symptomatic thromboembolic events | Up to 2 years
Treatment satisfaction (patient reported outcomes) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Multiple Locations, Algeria
- Multiple Locations, Egypt
- Multiple Locations, Indonesia
- Multiple Locations, Jordan
- Multiple Locations, Kazakhstan
- Multiple Locations, Kenya
- Multiple Locations, Kuwait
- Multiple Locations, Lebanon
- Multiple Locations, Malaysia
- Multiple Locations, Mexico
- Multiple Locations, Morocco
- Multiple Locations, Philippines
- Multiple Locations, Qatar
- Multiple Locations, Russia
- Multiple Locations, Saudi Arabia
- Multiple Locations, Singapore
- Multiple Locations, South Korea
- Multiple Locations, Taiwan
- Multiple Locations, Turkey (Türkiye)
- Multiple Locations, Ukraine
- Multiple Locations, United Arab Emirates